CLINICAL TRIAL: NCT03278041
Title: Effect of the Submental Artery Island Flap Versus Maxillary Obturator Prosthesis on the Quality of Life in Patients With Palatal Defects. (Randomized Controlled Clinical Study)
Brief Title: Effect of the Submental Artery Island Flap Versus Maxillary Obturator Prosthesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, OMAR ALADASH, Principle Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 454
Record Dates: First submitted 2017-09-07; First posted 2017-09-11 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Patient With Partial Maxillectomy; Submental Island Flap; Maxillary Obturator

STUDY DESIGN:
Masking Description: Because the two interventions used in this trial are clearly different and easly recognized by the participants and investigators, neither investigator AlAdashi O nor Participants can be blinded.
  Similarly, the Assessor (Participants) can't be blinded. The statistician will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- surgical reconstruction with submental flap (Experimental): surgical reconstruction with submental flap
  Interventions: Procedure: Submental flap for palatal reconstruction
- maxillary obturator (Active Comparator): maxillary obturator
  Interventions: Device: maxillary obturator

INTERVENTIONS:
Procedure: Submental flap for palatal reconstruction — Under General Anesthesia the tumor in the maxilla will be resected (partial maxillectomy) with a safety margin, then the defect will be reconstructed immediately by :
  Submental artery flap : from submental area with 1 cm distance from inferior mandibular border in paddle shape.
  * 1st step will be identify the facial artery and vein,
  * 2nd step dissection and extend toward midline in subplatsmal plane. The flap contains submental artery and vein.
  * 3rd step creating submucous tunnel between vestibular border of post maxillectomy defect and to extraoral incision .
  The flap will be through the oral cavity and will be anchored to the intact remaining hard plate with bone sutures by 2-0 vicryl® suture.
  Arms: surgical reconstruction with submental flap
Device: maxillary obturator — immediate surgical obturator
  Arms: maxillary obturator

SUMMARY:
The aim of the study is to compare maxillary obturator versus submental artery flap after partial maxillectomy in the aspect of Quality of life outcomes.

DETAILED DESCRIPTION:
The maxillary defects created by surgical removal of tumors result in communication between the oral and nasal cavities that in turn impair speech, swallowing, mastication, and facial esthetics, all of which consequently affect social behavior and quality of life (QoL). Consequently, the QoL need to be evaluated in patients with head and neck cancer because surgical resections and associated problems can affect QoL in significant ways.

University of Washington Head and Neck questionnaire is one of the measuring tools of the Quality of life, this UW-QOL questionnaire tests 12 domains relating to the patient with head and neck cancer. The sum score is calculated by adding together the scores for the 12 domains and dividing by 12 for a score from 0 (for poor health) to 100 (good health).

The maxillary defects reconstruction could be approached with prosthetic obturators rehabilitation or through surgical correction.

The obturator prostheses have many advantages that include; the easy visualization of the defect site, which allows for the detection of cancer recurrence; a reduction in the hospitalization period and costs; the ability to avoid a second operation; and the immediate re-establishment of facial morphology and oral functioning.However, several disadvantages to the maxillary obturator exist, including the discomfort of wearing a prosthesis, the inconvenience of removing and cleaning the prosthesis, the inability to successfully retain a prosthesis when the defect is large or when dentition is lacking, and the frequent need for readjustments by a prosthodontist.

The surgical intervention could be with various approaches that provide the reconstruction of communication and yields good results for the reconstruction of small defects.

The most commonly used surgical technique is the free tissue transfers that associated with increased hospital time and flap donor area morbidity. Nonetheless, Study conducted by Rogers et al., compared obturator prosthesis versus free flap surgical repair of the maxillary defect, the result revealed that there were no statistically significant differences were found between the two groups regarding quality of life measured with UW-QOL, although there was a tendency for obturator patients to indicate more problems with appearance. In this study, the obturator group recorded UW-QOL mean of 74±8.

The drawbacks of previous techniques have led to a search for alternate solutions, the use of a pedicle submental artery island flap is introduced as a new surgical option for head and neck tumor reconstruction. The advantages of this approach coming from its donor site can be performed in very thin section, pliability, and versatility in design. Moreover, the submental flap can be easily raised and involves shorter operative and hospital time compared to the free-flap procedure.

The pedicle submental artery island flap can be an excellent choice in patients with a high American Society of Anesthesiologists (ASA) risk score; moreover, this modality is effective in elderly patients, where the potential complications linked to microsurgical procedures are avoided.

There is no published study until now comparing pedicle submental artery island flap with prosthetic obturators. So that the aim of this study is to answer the following question "After partial maxillectomy in patients with a palatal defect, Does the submental artery flap offer different effect on the improvement of the quality of life when compared to maxillary obturator?"

ELIGIBILITY:
Inclusion Criteria:

All subjects were required:

1. All patients suffering from midface defects that involving palatal-maxillary bone are included.
2. All ages and both sexes were included in this study.
3. Patients with good general condition allowing major surgical procedure under general anesthesia.
4. Be physically and psychologically able to tolerate procedures.
5. Be cooperative to return for follow-up, examinations and evaluation.

Exclusion Criteria:

1. Patient who physically and psychologically not able to tolerate procedures. Because they cannot able to tolerate procedures and may discontinue the follow-up visits.
2. Be Uncooperative to return for follow-up, examinations and evaluation.
3. Patients with any systemic disease (e.g uncontrolled diabetic, bisphosphonates …..ect) because that may affect normal healing.
4. Patient with bad oral hygiene.Because poor oral hygiene can cause inflammation which induces pain that effect outcome reading.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-01-30 (Estimated); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-01-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life | one months post operative
  measured by University of Washington Head and Neck questionnaire(UW-QOL).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry-cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided